CLINICAL TRIAL: NCT02973919
Title: EMDR in Spider Phobia: Work Mechanisms and Treatment Outcome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Regensburg (Other)
Responsible Party: Principal Investigator, Shiban Youssef, Phd, University of Regensburg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: URegensburg
Record Dates: First submitted 2016-11-14; First posted 2016-11-28 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-11

CONDITIONS: Spider Phobia
MeSH Terms: conditions — Arachnophobia | interventions — Virtual Reality Exposure Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Eye movements (Experimental): Eye Movement Desensitization and Reprocessing Therapy + virtual reality exposure therapy
  Interventions: Behavioral: Eye Movement Desensitization and Reprocessing Therapy; Behavioral: Virtual Reality Exposure Therapy
- Control (Active Comparator): virtual reality exposure therapy
  Interventions: Behavioral: Virtual Reality Exposure Therapy

INTERVENTIONS:
Behavioral: Eye Movement Desensitization and Reprocessing Therapy — In 1989, Shapiro discovered that while talking about negative life events or thoughts, rhythmic eye movements on a horizontal axis can alleviate the associated vividness and burden (Shapiro, 1989). She established the psychodynamic-behavioral Eye Movement Desensitization and Reprocessing (EMDR) Therapy, which includes the induction of rhythmic eye movements as a central feature. EMDR is regarded as an efficient treatment tool. Several times it has also been successfully applied in the field of specific phobias (de Jongh, ten Broeke, & Renssen, 1999; de Jongh, Holmshaw, Carswell, & van Wijk, 2011; Lapsekili & Yelboga, 2014; Muris, Merckelbach, van Haaften, & Mayer, 1997) and there is a standard protocol for using EMDR on specific fears and phobias (de Jongh, 2015).
  Arms: Eye movements
Behavioral: Virtual Reality Exposure Therapy — Exposure to fear-evoking stimuli is conducted more often in virtual environments using simulators or similar computer-technologies (Virtual Reality Exposure Therapy, VRET). One great advantage of using VR-technologies is that it is possible to create an environment which is highly controllable by its creators. Feared stimuli or scenarios can be varied on individual purposes and presented several times. This facili- tates the practice of exposure-based treatments especially for situations or places diffi- cult to access or requiring a considerable amount of time and/or money (e.g. being in war zones or a passenger on a flight), where in vivo exposures have often not been con- ducted or only in a limited manner (Mühlberger & Pauli, 2011).

SUMMARY:
The goal of this study is to increase the efficiency of exposure in virtual reality (VR).

Based on the EMDR research the investigators would like to show that the implementation of eye movements during the VR exposure results in a faster physiological relaxation response among probands with spider phobia, which has a positive effect on the subjective and behavioral efficacy of the VR exposure.

DETAILED DESCRIPTION:
The VR paradigm consists of one room with a spider in it. The proband is supposed to look at it for a few minutes. This exposure is repeated several times.

In the experimental group a ball appears during the exposure, that moves horizontally across the room. The probands are supposed to follow this movement with their eyes.

EDA, EKG and respiration are being recorded. Furthermore the subjective and behavioral spider phobia is measured before, during and after the exposure to determine occurring changes.

ELIGIBILITY:
Inclusion Criteria:

* the Structured Clinical Interview for DSM-IV (SCID, First et al., 2002; applied German translation: Strukturiertes Klinisches Interview für DSM-IV, Achse I, SKID I, Wittchen et al., 1997), in order to get a reliable diagnosis of spider phobia

Exclusion Criteria:

* pregnancy
* current psychopharmacological medication
* current involvement in psychiatric- or psychotherapeutic treatment
* cardiovascular or neurological diseases
* color blindness
* hearing disorders

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2015-07; Primary Completion 2015-12 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Change in Behavioral Assessment Test (BAT) in vivo | 5 minutes before, 5 minutes after intervention and during folow up (2 weeks post Intervention)
  expected fear just before getting started and actually present fear just before finishing

SECONDARY OUTCOMES:
Skin Conductance Reactivity (SCR) | during the VR-session
Electrocardiogram (ECG) | during the VR-session
  providing the Heart Rate (HR)
manipulation check electrode below the right eye (M. orbicularis oculi) | during the VR- exposure sessions (5 min x 4 sessions)
  for registering eye movements
Change in Subjective Fear Ratings | 1 min before and during ( each minute) exposure in Virtual Reality
  Subjective Units of Disturbance Scale

IPD SHARING:
Plan to Share IPD: No